CLINICAL TRIAL: NCT02245412
Title: A Phase 2A Study of ALXN1007 in Subjects With Newly Diagnosed Acute Graft-Versus-Host Disease Involving the Lower Gastrointestinal Tract
Brief Title: A Phase 2A Study of ALXN1007 in Participants With Newly Diagnosed Acute Lower Gastrointestinal Graft-Versus-Host Disease
Acronym: GIGVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early at the Sponsor's discretion, not due to safety concerns.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1007-GIGVHD-201
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Acute Graft-Versus-Host Disease; GIGVHD
Keywords: GIGVHD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ALXN1007 10 mg/kg once weekly (Experimental): Cohort 1, the first dosing cohort, received 10 mg/kg ALXN1007 IV once weekly for 8 weeks.
  Interventions: Biological: ALXN1007 10 mg/kg once weekly
- ALXN1007 20 mg/kg once weekly (Experimental): Cohort 2 received 20 mg/kg ALXN1007 IV once weekly for 8 weeks. For the first 2 participants enrolled, the first ALXN1007 dose was not to be administered on the same day and a safety and tolerability review was to take place after the second (and prior to the third) ALXN1007 dose for each participant. If the ALXN1007 dose was determined to be sufficiently tolerated by the participant, dosing was to continue for that participant. For any other participants enrolled in the dosing cohort, participants were not to proceed to the third ALXN1007 dose prior to the completion of the safety and tolerability review (of the first 2 doses) for the first 2 participants.
  Interventions: Biological: ALXN1007 20 mg/kg once weekly
- ALXN1007 20 mg/kg twice weekly (Experimental): Cohort 3 received 20 mg/kg ALXN1007 IV twice weekly for 8 weeks. For the first 2 participants enrolled, the first ALXN1007 dose was not to be administered on the same day and a safety and tolerability review was to take place after the second (and prior to the third) ALXN1007 dose for each participant. If the ALXN1007 dose was determined to be sufficiently tolerated by the participant, dosing was to continue for that participant. For any other participants enrolled in the dosing cohort, participants were not to proceed to the third ALXN1007 dose prior to the completion of the safety and tolerability review (of the first 2 doses) for the first 2 participants.
  Interventions: Biological: ALXN1007 20 mg/kg twice weekly

INTERVENTIONS:
Biological: ALXN1007 10 mg/kg once weekly — ALXN1007 is a recombinant humanized monoclonal antibody that binds to complement component C5a and its metabolite C5a desArg.
  Arms: ALXN1007 10 mg/kg once weekly
Biological: ALXN1007 20 mg/kg once weekly — ALXN1007 is a recombinant humanized monoclonal antibody that binds to complement component C5a and its metabolite C5a desArg.
  Arms: ALXN1007 20 mg/kg once weekly
Biological: ALXN1007 20 mg/kg twice weekly — ALXN1007 is a recombinant humanized monoclonal antibody that binds to complement component C5a and its metabolite C5a desArg.
  Arms: ALXN1007 20 mg/kg twice weekly

SUMMARY:
The objectives of this trial were to evaluate the safety, tolerability, pharmacokinetics/pharmacodynamics (PK/PD) and efficacy of intravenous (IV) ALXN1007 in participants with acute graft-versus-host disease (GVHD) of the lower gastrointestinal (GI) tract.

DETAILED DESCRIPTION:
This was a Phase 2A open-label, non-randomized study to evaluate the safety, tolerability, PK/PD, and efficacy of ALXN1007 (a C5a inhibitor) in up to 36 participants with newly diagnosed acute GVHD of the lower GI tract. All participants meeting the inclusion and exclusion criteria for the study were to receive ALXN1007 over an 8 week treatment period. Participants in Cohort 1, the first dosing cohort, were to receive 10 milligrams/kilogram (mg/kg) ALXN1007 administered IV once weekly for 8 weeks. Participants in Cohort 2 were to receive 20 mg/kg ALXN1007 IV once weekly for 8 weeks. Participants in Cohort 3 were to receive 20 mg/kg ALXN1007 IV twice weekly for 8 weeks. All doses of ALXN1007 were to be administered as a continuous IV infusion.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be males or females age 18 years or older.
* Participants with Stage 1 to 4 (per the Modified Keystone Grading Schema) acute GVHD of the lower GI tract, without signs of chronic GVHD, at the time of diagnosis, which developed in the first 180 days following allogeneic hematopoietic cell transplantation (HCT) using bone marrow, peripheral blood, or cord blood; or after preplanned donor lymphocyte infusion.
* Participants are willing to undergo or must have had an endoscopy of the upper and/or lower GI tract and biopsy to confirm GI GVHD.
* Participants must be receiving systemic corticosteroids.
* Participants with an absolute neutrophil count (ANC) >500/microliter (μL) at Screening.
* Participants and spouse/partner who are of childbearing potential must be using high effective contraception consisting of 2 forms of birth control (at least 1 of which much be barrier method) starting at Screening and continuing through the entire study (for at least 3 months after the last dose of ALXN1007 if study treatment is stopped early or participant withdraws consent).
* Male participants must not donate sperm during the Screening and Treatment periods, and for at least 3 months after the last dose of ALXN1007.

  * Stage of acute GVHD of the lower GI tract will be determined using the Modified Keystone Grading Schema.

Exclusion Criteria:

* Participants with a body weight > 140 kg (for Cohorts dosing 20 mg/kg of ALXN1007 and higher only).
* Participants with signs and symptoms of chronic GVHD.
* Participants with an active uncontrolled infection.
* Participants who test positive for Clostridium difficile (C. difficile) at Screening.
* Participants with relapsed/persistent malignancy requiring rapid immune suppression withdrawal.
* Participants who received an unplanned (not part of the original transplant therapy plan) donor lymphocyte infusion.
* Participants who received previous systemic treatment for acute GVHD, except for a maximum of 3 days (72 hours) of 2 mg/kg corticosteroid therapy.
* Participants with unresolved veno-occlusive disease of the liver.
* Participants with creatinine clearance <40 milliliters (mL)/minute at Screening, as calculated by the Cockcroft-Gault formula.
* Participants known to be infected with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* Participants known to have an uncontrolled thyroid disorder.
* Participants who are pregnant, breast feeding, or sexually active and unwilling to use effective birth control for the duration of the study.
* Participants who participated in any other investigational drug trial or had exposure to any other investigational agent, device, or procedure <4 weeks prior to Screening and throughout the entire trial, with the exception of investigational drugs administered prophylactically for cytomegalovirus (CMV) post allogeneic HCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (9):
  - City of Hope, Duarte, California
  - Emory University Hospital, Atlanta, Georgia
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Medicine - Hematology, Oncology and Transplantation Office, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Abramson Cancer Perelman Center for Advanced Medicine, University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- France (3):
  - CHU de Grenoble - Hôpital Nord, Grenoble, Isere
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - Centre François, Gironde
  - Hôpital Saint-Louis, Paris

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants with newly diagnosed acute graft-versus-host disease (GVHD) of the lower gastrointestinal (GI) tract.
Groups:
- ALXN1007 10 mg/kg Once Weekly: Cohort 1, the first dosing cohort, received 10 milligrams/kilogram (mg/kg) ALXN1007 intravenously (IV) once weekly for 8 weeks.
Period: Treatment Period
Arm/Group | ALXN1007 10 mg/kg Once Weekly | ALXN1007 20 mg/kg Once Weekly | ALXN1007 20 mg/kg Twice Weekly
Started | 17 | 6 | 2
Received at Least 1 Dose of Study Drug | 17 | 6 | 2
Modified Full Analysis Set (mFAS) (The mFAS included all participants who had at least 1 dose of ALXN1007 and had GI GVHD confirmed.) | 16 | 6 | 2
Completed | 12 | 3 | 2
Not Completed | 5 | 3 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Biopsy did not confirm GI GVHD | 1 | 0 | 0
Period: Follow-Up Period
Arm/Group | ALXN1007 10 mg/kg Once Weekly | ALXN1007 20 mg/kg Once Weekly | ALXN1007 20 mg/kg Twice Weekly
Started | 13 (One participant who discontinued Study Drug in Treatment Period continued to Follow-Up Period.) | 4 (One participant who discontinued Study Drug in Treatment Period continued to Follow-Up Period.) | 2
Completed | 8 | 2 | 0
Not Completed | 5 | 2 | 2
Not completed — Death | 4 | 2 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Other - Terminated by Sponsor | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of ALXN1007.
Groups:
- Total: Total of all reporting groups
Arm/Group | ALXN1007 10 mg/kg Once Weekly | ALXN1007 20 mg/kg Once Weekly | ALXN1007 20 mg/kg Twice Weekly | Total
Number analyzed (Participants) | 17 | 6 | 2 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (14.27) | 47.7 (13.14) | 70.5 (2.12) | 54.2 (14.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 1 | 11
  Male | 9 | 4 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 14 | 5 | 2 | 21
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 16 | 3 | 2 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 6 | 2 | 24
  France | 1 | 0 | 0 | 1
Acute GVHD Staging [Count of Participants; unit: Participants] — The Modified Keystone Grading Schema: Skin - Stage 0 = No Rash, Stage 1 = Rash <25% body surface area (BSA), Stage 2 = 25% to 50% BSA, Stage 3 = >50% BSA, Stage 4 = bullae and desquamation; Lower GI Tract (determining stool volume over a 24-hour period) - Stage 0 = <500 milliliters (mL), Stage 1 = 500 to 1000 mL, Stage 2 = 1001 to 1500 mL, Stage 3 = >1500 mL, Stage 4 = severe abdominal pain +/- ileus, frank blood, or melena; Liver (bilirubin levels) - Stage 0 = ≤2 mg/deciliter (dL), Stage 1 = 2.1 to 3 mg/dL, Stage 2 = 3.1 to 6 mg/dL, Stage 3 = 6.1 to 15 mg/dL, and Stage 4 = >15 mg/dL.
  Participants
    Skin: Staging Score 0 | 14 | 6 | 1 | 21
    Skin: Staging Score 1 | 0 | 0 | 0 | 0
    Skin: Staging Score 2 | 3 | 0 | 1 | 4
    Skin: Staging Score 3 | 0 | 0 | 0 | 0
    Skin: Staging Score 4 | 0 | 0 | 0 | 0
    Lower GI Tract: Staging Score 0 | 7 | 0 | 0 | 7
    Lower GI Tract: Staging Score 1 | 4 | 1 | 1 | 6
    Lower GI Tract: Staging Score 2 | 1 | 3 | 0 | 4
    Lower GI Tract: Staging Score 3 | 5 | 1 | 1 | 7
    Lower GI Tract: Staging Score 4 | 0 | 1 | 0 | 1
    Liver: Staging Score 0 | 17 | 6 | 2 | 25
    Liver: Staging Score 1 | 0 | 0 | 0 | 0
    Liver: Staging Score 2 | 0 | 0 | 0 | 0
    Liver: Staging Score 3 | 0 | 0 | 0 | 0
    Liver: Staging Score 4 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Acute Graft-Versus-Host Disease (GVHD) Response Rate At Day 28
Description: The number of participants with overall acute GVHD response was determined at Day 28. Acute Overall GVHD is defined as improvement from diagnosis in any organ by at least 1 stage, without progression in any other organ, and with no additional therapy being administered. Acute GVHD staging included skin, liver, and GI assessments, which were to be performed using the Modified Keystone Grading Schema. Deaths were considered nonresponders; otherwise last postbaseline values were carried forward for imputation of missing responses. Modified Keystone Grading Schema: Skin - Stages 0 = No Rash, 1 = Rash <25% body surface area (BSA), 2 = 25% to 50% BSA, 3 = >50% BSA, 4 = bullae, desquamation; Lower GI Tract (stool volume over 24 hours) - Stages 0 = <500 mL, 1 = 500 to 1000 mL, 2 = 1001 to 1500 mL, 3 = >1500 mL, 4 = severe abdominal pain +/- ileus, frank blood, or melena; Liver (bilirubin levels) - Stages 0 = ≤2 mg/dL, 1 = 2.1 to 3 mg/dL, 2 = 3.1 to 6 mg/dL, 3 = 6.1 to 15 mg/dL, 4 = >15 mg/dL.
Time Frame: Day 28
Population: Participants in the mFAS Population - In the 10 mg/kg ALXN1007 once weekly dose group, 1 participant was prematurely discontinued after receiving a single dose due to lack of confirmed GI GVHD.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1007 10 mg/kg Once Weekly | ALXN1007 20 mg/kg Once Weekly | ALXN1007 20 mg/kg Twice Weekly
Number analyzed (Participants) | 16 | 6 | 2
Participants | 10 | 3 | 1

2. Secondary Outcome: Pharmacokinetics (PK): Time To Maximum Observed Concentration In Plasma (Tmax) Of IV ALXN1007
Description: The Tmax of ALXN1007 was measured on Treatment Days 1, 28, and 49, from blood samples collected at time points relative to the dosing of ALXN1007. PK assessments were to have been measured from Baseline, Treatment Days 7, 14, 21, 28, 35, 42, 49, 56, and Follow-up Days 86, 180, and Early Termination (ET).
  Due to the early termination of the study and the clinical development of the ALXN1007 program, a number of PK analyses were not completed. PK data for the 20 mg/kg ALXN1007 once weekly dosing group and the 20 mg/kg ALXN1007 twice weekly dosing group are not available.
Time Frame: Predose up to 72 hours postdose
Population: PK population: All participants in the 10 mg/kg ALXN1007 once weekly dose group who received at least 1 dose of ALXN1007 and who had evaluable PK and pharmacodynamic (PD) data.
Measure: Median (Full Range); unit: hours
Arm/Group | ALXN1007 10 mg/kg Once Weekly | ALXN1007 20 mg/kg Once Weekly | ALXN1007 20 mg/kg Twice Weekly
Number analyzed (Participants) | 10 | 0 | 0
hours
  Tmax Day 1 | 1.033 [0.983 to 5.0] |  |
  Tmax Day 28 | 1.03 [1.0 to 5.0] |  |
  Tmax Day 49 | 1.25 [1.0 to 1.8] |  |

3. Secondary Outcome: PK: Maximum Observed Concentration In Plasma (Cmax) Of IV ALXN1007
Description: The Cmax of ALXN1007 was measured on Treatment Days 1, 28, and 49, from blood samples collected at time points relative to the dosing of ALXN1007. PK assessments were to have been measured from Baseline, Treatment Days 7, 14, 21, 28, 35, 42, 49, 56, and Follow-up Days 86, 180, and Early Termination (ET).
  Due to the early termination of the study and the clinical development of the ALXN1007 program, a number of PK analyses were not completed. PK data for the 20 mg/kg ALXN1007 once weekly dosing group and the 20 mg/kg ALXN1007 twice weekly dosing group are not available.
Time Frame: Predose up to 72 hours postdose
Population: PK population: All participants in the 10 mg/kg ALXN1007 once weekly dose group who received at least 1 dose of ALXN1007 and who had evaluable PK and PD data.
Measure: Median (Full Range); unit: ug/mL
Arm/Group | ALXN1007 10 mg/kg Once Weekly | ALXN1007 20 mg/kg Once Weekly | ALXN1007 20 mg/kg Twice Weekly
Number analyzed (Participants) | 10 | 0 | 0
ug/mL
  Cmax Day 1 | 270 [156 to 318] |  |
  Cmax Day 28 | 383 [283 to 409] |  |
  Cmax Day 49 | 421 [207 to 450] |  |

4. Secondary Outcome: PK: Area Under The Plasma (Or Serum) Concentration Versus Time Curve (AUC) Of IV ALXN1007
Description: The AUC of ALXN1007 was measured on Treatment Days 1, 28, and 49, from blood samples collected at time points relative to the dosing of ALXN1007. PK assessments were to have been measured from Baseline, Treatment Days 7, 14, 21, 28, 35, 42, 49, 56, and Follow-up Days 86, 180, and Early Termination (ET).
  Due to the early termination of the study and the clinical development of the ALXN1007 program, a number of PK analyses were not completed. PK data for the 20 mg/kg ALXN1007 once weekly dosing group and the 20 mg/kg ALXN1007 twice weekly dosing group are not available.
Time Frame: Predose up to 72 hours postdose
Population: as for outcome 3
Measure: Median (Full Range); unit: h*ug/mL
Arm/Group | ALXN1007 10 mg/kg Once Weekly | ALXN1007 20 mg/kg Once Weekly | ALXN1007 20 mg/kg Twice Weekly
Number analyzed (Participants) | 10 | 0 | 0
h*ug/mL
  AUC Day 1 | 13079 [7429 to 20113] |  |
  AUC Day 28 | 34957 [22432 to 50439] |  |
  AUC Day 49 | 41919 [17182 to 59625] |  |

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Adverse Events were reported for the mFAS, which included all participants who received at least 1 dose of ALXN1007 and for whom GI GVHD was confirmed through biopsy.
Arm/Group | ALXN1007 10 mg/kg Once Weekly | ALXN1007 20 mg/kg Once Weekly | ALXN1007 20 mg/kg Twice Weekly
All-Cause Mortality (participants affected / at risk) | 6/17 | 3/6 | 1/2
Serious Adverse Events (participants affected / at risk) | 13/17 | 4/6 | 2/2
Other Adverse Events (participants affected / at risk) | 17/17 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN1007 10 mg/kg Once Weekly (N=17) | ALXN1007 20 mg/kg Once Weekly (N=6) | ALXN1007 20 mg/kg Twice Weekly (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Graft versus host disease (Immune system disorders) | 0 | 1 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 4 | 2 | 2
BK virus infection (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 11 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Precursor B-lymphoblastic lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN1007 10 mg/kg Once Weekly (N=17) | ALXN1007 20 mg/kg Once Weekly (N=6) | ALXN1007 20 mg/kg Twice Weekly (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Eyelid margin crusting (Eye disorders) | 1 | 0 | 0
Scleral hyperaemia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Vitreous degeneration (Eye disorders) | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Device related thrombosis (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1
Oedema (General disorders) | 2 | 1 | 0
Oedema peripheral (General disorders) | 7 | 2 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Graft versus host disease in skin (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1 | 1
Adenovirus infection (Infections and infestations) | 1 | 1 | 0
BK virus infection (Infections and infestations) | 1 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Colitis herpes (Infections and infestations) | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Enterococcal infection (Infections and infestations) | 2 | 1 | 0
Epstein-Barr viraemia (Infections and infestations) | 0 | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 2 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Human herpesvirus 6 infection (Infections and infestations) | 2 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Rotavirus infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0
Blood immunoglobulin G decreased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 2 | 0
White blood cell count decreased (Investigations) | 1 | 3 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Akathisia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Tardive dyskinesia (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Depressive symptom (Psychiatric disorders) | 1 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Cystitis viral (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication rights are tied to the completion of the multi-center publication

DOCUMENTS (2):
  • Study Protocol (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT02245412/Prot_002.pdf
  • Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT02245412/SAP_003.pdf